CLINICAL TRIAL: NCT03975049
Title: A Prospectively Randomized Phase III Trial Comparing Short-term mFOLFOXIRI, Long-term mFOLFOX6 and Traditional Chemoradiation as Preoperative Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: Triplet Combination or Doublet Regimen Versus Chemoradiation as Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO201
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Rectal Cancer; Chemotherapy Effect
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; FOLFOXIRI protocol; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5-Fu + RT (Active Comparator): 5Fu + RT for five weeks --- 6-8 weeks of interval --- TME --- mFOLFOX * 6-8
  Interventions: Radiation: Chemoradiation
- mFOLFOXIRI (Experimental): mFOLFOXIRI * 4 --- TME --- mFOLFOXIRI * 4
  Interventions: Drug: FOLFOXIRI Protocol
- mFOLFOX (Experimental): mFOLFOX * 9 --- TME --- mFOLFOX * 3
  Interventions: Drug: Folfox Protocol

INTERVENTIONS:
Radiation: Chemoradiation — Fluorouracil 225 mg/m2/day continuous intravenous infusion on weekdays for five weeks; local irradiation 2GY/day on weekdays, totally 50GY.
  Arms: 5-Fu + RT
Drug: FOLFOXIRI Protocol — Oxaliplatin 85 mg/m2 on day 1; irinotecan 150 mg/m2 on day 1; leucovorin 400 mg/m2 on day 1; fluorouracil 2400 mg/m2 civ over 46h; treatment will be repeated every 14 days; prophylactic G-CSF support is recommended.
  Arms: mFOLFOXIRI
Drug: Folfox Protocol — Oxaliplatin 85 mg/m2 on day 1; leucovorin 400 mg/m2 on day 1; fluorouracil 400 mg/m2 bolus and 2400 mg/m2 civ over 46h; treatment will be repeated every 14 days.
  Arms: mFOLFOX

SUMMARY:
Preoperative radiation with single agent chemotherapy as sensitizer is the standard care of locally advanced rectal cancer.

Local irradiation significantly increases surgical complications and impairs quality of life.

Combination chemotherapy alone seems promising and provides similar benefit to chemoradiation as neoadjuvant therapy.

Early administration of systemic therapy is also proved beneficial for long-term survival.

The purpose of this study is to compare the efficacy of chemotherapy alone with short-term modified FOLFOXIRI or long-term mFOLFOX with standard chemoradiation as neoadjuvant therapy for locally advanced rectal cancer.

DETAILED DESCRIPTION:
Patients with cT3-4 or cN+ and cM0 by pelvic MR and chest + abdominal CT scan will be randomized to the following three groups:

Group A: Traditional chemoradiation.

Fluorouracil 225 mg/m2/day continuous intravenous infusion on weekdays for five weeks; local irradiation 2GY/day on weekdays, totally 50GY.

At the end of chemoradiation, patients will receive an evaluation with MR and CT scan.

If the efficacy is defined as CR, PR or SD, the TME will be performed in 6-8 weeks since the last irradiation.

If the disease progress with the possibility of R0 resection, the operation will be given soon.

If the tumor progress to impossible for R0 resection, the salvage chemotherapy will be given accordingly.

Adjuvant chemotherapy of 6-8 cycles of mFOLFOX will be administered 3-4 weeks after R0 resection.

Group B: Short-term mFOLFOXIRI.

Oxaliplatin 85 mg/m2 on day 1; irinotecan 150 mg/m2 on day 1; leucovorin 400 mg/m2 on day 1; fluorouracil 2400 mg/m2 civ over 46h; treatment will be repeated every 14 days; prophylactic G-CSF support is recommended.

Patients are planned to receive 4 cycles of mFOLFOXIRI regimen preoperatively and postoperatively, respectively.

Before operation, efficacy evaluations will be performed every two cycles by CT and MR scan.

If the evaluation is defined as no progression without severe toxicity, the next 2 cycles will be given.

If the primary lesion progress without distant metastasis, patients will be assigned to group A.

If distant metastasis occurr during chemotherapy, patients will withdraw from the trial and be treated further at the discretion of attending physicians.

Postoperative chemotherapy will initiate 3-4 weeks after R0 resection.

Group C: Long-term mFOLFOX.

Oxaliplatin 85 mg/m2 on day 1; leucovorin 400 mg/m2 on day 1; fluorouracil 400 mg/m2 bolus and 2400 mg/m2 civ over 46h; treatment will be repeated every 14 days.

Patients are planned to receive 8-9 cycles of mFOLFOX regimen preoperatively and 3-4 cycles postoperatively.

Efficacy evaluations will be performed every three cycles by CT and MR scan before TME.

If the evaluation is defined as no progression without severe toxicity, the next 3 cycles of mFOLFOX will be given with the maximum of 9 cyces.

If the primary lesion progress without distant metastasis, patients will be assigned to group A.

If distant metastasis occurr during chemotherapy, patients will withdraw from the trial and be treated further at the discretion of attending physicians.

Postoperative chemotherapy will initiate 3-4 weeks after R0 resection.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age: 18 to 75 years old;
* 2）Histological diagnosis of rectal adenocarcinoma;
* 3）Distance form anal margin ≤ 12cm: cT3-4 or cN+ and cM0 by pelvic MR and chest + abdominal CT, estimated possible for R0 resection;
* 4）There is no signs of intestinal obstruction, or obstruction of intestinal after treating with proximal colostomy has been relieved;
* 5）Patients did not previously receive rectal surgery, chemotherapy or radiation therapy , biological treatment , except for endocrine therapy;
* 6）ECOG Performance Status :0-1
* 7）Life expectancy: more than 3 years;
* 8）sufficient bone marrow, liver and kidney function.

Exclusion Criteria:

* 1）Arrhythmia requires treatment with antiarrhythmia (except for beta-blockers or digoxin), symptomatic coronary artery disease, myocardial ischemia (myocardial infarction within the last 6 months) or congestive heart failure exceeding NYHA class II;
* 2）Severe hypertension with poor control;
* 3）History of HIV infection or active phase of chronic hepatitis B or C infection with high copy viral DNA;
* 4）Other active serious infections according to NCI-CTC version 4.0;
* 5）There is preoperative evidence for distant metastasis outside pelvis;
* 6）Cachexia and organ function decompensation
* 7）History of pelvic or abdominal radiotherapy;
* 8）Multiple primary cancer;
* 9）Patients with epilepcy requiring treatment ( steroids or antiepileptic treatment);
* 10）History of other malignant tumors within 5 years, except for cured cervical carcinoma in situ or skin basal cell carcinoma;
* 11）Drug abuse and medical, psychological or social conditions interfering patient participation in research or the evaluation of research results;
* 12）Any allergy to clinical research drugs or any drugs associated with this study;
* 13）Any unstable condition or condition that may endanger safety and compliance of patients;
* 14）Pregnancy or the lactating female without adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years
  The interval from randomization to local recurrence, distant metastasis, death or the last follow-up.

SECONDARY OUTCOMES:
Recurrence-free survival | 3 years
  The interval from randomization to local recurrence, death or the last follow-up.
Metastasis-free survival | 3 years
  The interval from randomization to distant metastasis, death or the last follow-up.
Surgical complication | 3 years
  Surgical complication including anastomotic leakage, anastomotic stricture, intestinal obstruction, postoperative pelvic bleeding and poor wound healing.
Treatment related quality of life | up to 3 years
  EORTC QOL questionaire

OTHER OUTCOMES:
Tumor regression grade after neoadjuvant therapy | 3 months
  According to pathological slides

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No